CLINICAL TRIAL: NCT00696943
Title: An Open-label, Multi-center Study to Evaluate [18F]-ML-10 as a PET Imaging Radiotracer for Early Detection of Response of Brain Metastases to Stereotactic Radio Surgery (SRS)
Brief Title: 18F ML-10 for Early Detection of Response of Brain Metastases to SRS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Replaced by a global study protocol NST-CA004
Sponsor: Aposense Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NST-CA005CTIL
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2008-11

CONDITIONS: Metastasis to Brain of Unknown Primary
Keywords: cell death; PET imaging; brain metastases; stereotactic radiosurgery
MeSH Terms: conditions — Brain Neoplasms | interventions — 5-fluoropentyl-2-methylmalonic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F-ML-10, (Experimental): Pre-treatment baseline and post treatment follow-up 18F ML-10 PET/CT sessions.
  Interventions: Drug: ([18F]-ML-10)

INTERVENTIONS:
Drug: ([18F]-ML-10) — [18F]-ML-10 was administered as an intravenous bolus injection (in 3-10 ml sterile saline solution, containing no more than 10% ethanol by volume). The radiation dose of [18F]-ML-10 administered at each session was 300-500 MBq (8.1-13.5 mCi).
  Other Names: 2-(5-fluoro-pentyl)-2-methyl-malonic-acid

SUMMARY:
The purpose of this study is to evaluate the potential of [18F]-ML-10 to serve as a non-invasive imaging tool for the early detection of apoptosis in brain metastases in response to radiation therapy, in patients subjected to stereotactic radiosurgery (SRS). Such early detection may improve clinical management of patients with brain metastases, as it may help early identification of non-responders, and subsequently potentially lead to optimization of radiation techniques such as the need for whole brain radiation therapy (WBRT), addition of brain penetrating chemotherapy or an early decision on referral of the patient with non-responsive lesions to surgery or to systemic chemotherapy. The experimental design of the present study aims to evaluate the potential of non-invasive PET examination with [18F]-ML-10, to provide the clinician with an assessment of response early in the course of treatment, via non-invasive molecular imaging of radiation-induced apoptosis. This information on tumor responsiveness is currently available only several weeks to months after completion of radiotherapy.

DETAILED DESCRIPTION:
Early assessment of the efficacy of anti-cancer therapy is highly desirable and an unmet need in clinical oncology. Currently, treatment efficacy is mostly measured by following tumor size by anatomical imaging (CT scan or MRI). However, changes in tumor size may be observed only after several weeks to several months after completion of treatment. Meanwhile, in cases where there is no response, the patient is unnecessarily exposed to treatment's side effects, and precious time may be lost before the initiation of an alternative, potentially more beneficial line of therapy. Therefore, there is an urgent and serious need for better tools for monitoring of tumor response to anti-cancer treatments.

To address this need, [18F]-ML-10, a novel small molecular-weight probe (MW 205) was developed for clinical detection of apoptosis in vivo by positron emission tomography (PET). [18F]-ML-10 is a member of the ApoSense family of compounds, a novel class of molecular probes for molecular imaging of cell death. The first clinical indication for which [18F]-ML-10 is being developed is imaging of apoptosis in clinical oncology to monitor tumor response to radiation therapy.

Previous preclinical and clinical studies have substantiated the safety of [18F]-ML-10, its very high stability in vivo, its favorable biodistribution profile, and its efficacy in clinical detection of cell death. In preclinical studies, the selective retention of [18F]-ML-10 in the focus of the neurovascular cell death in cerebral ischemia was demonstrated in respective animal models. [18F]-ML-10 has been examined in two clinical trials in Uppsala Imanet, Sweden, and has been found safe in administration to healthy subjects and to elderly subjects with acute ischemic cerebral stroke. In these clinical trials, [18F]-ML-10 was also found efficacious in the clinical imaging of apoptosis, being either physiological apoptosis as observed in the testes in young healthy males, and pathological cell death, as observed in the brains of patients with acute ischemic cerebral stroke.

ELIGIBILITY:
Inclusion Criteria:

The Patient may only be included in the study if ALL of the following statements are fulfilled:

1. Male or female patient diagnosed with metastatic non hematological cancer, with up to 4 brain metastases of which at least one has a minimal diameter of 1.5cm , as assessed by MRI (utilized for SRS planning) and is scheduled for SRS. These metastases will be defined as target lesions.
2. Patient is ≥ 18 years of age at the time of signature of the informed consent form.
3. Fully conscious patient who has been given written and verbal information, and has then provided an informed consent.
4. Patient who is able to cooperate with the studies requirements to lie still during PET/CT imaging scans, which may last for up to 3 hours.
5. ECOG performance status of 0, 1 or 2 at the time of enrollment.
6. Patient with life expectancy ≥ 12 weeks.
7. Adequate renal function and adequate hepatic function as assessed by standard laboratory criteria and defined as:

   1. Creatinine clearance ≥ 60 ml/min/1.73m2according to Cockroft & Gault Formula
   2. Total bilirubin ≤ 1.5 times the ULN
   3. Aspargine aminotransferase (AST), alanine aminotransferase (ALT) ≤ 3 times the ULN in patients without liver metastases; ≤ 5 times the ULN in patients with liver metastases
8. Serum calcium levels, adjusted to albumin level, within normal limits.
9. For a female patient, pregnancy or breast-feeding are restricted. Woman of child bearing potential must have a negative serum pregnancy test at screening.

Exclusion Criteria:

If any apply, the patient must not be included in the study:

1. Unstable medical condition, such as severe ischemic heart disease, liver disease or pulmonary disease, which may risk the patient during the study, as judged by the investigator.
2. Any indication of imminent brain herniation
3. Any known psychiatric disorder other than mild depression or anxiety.
4. Known allergy to Gadolinium
5. Other condition that might jeopardize the safety of the patient or the evaluation of the study results, as judged by the investigator.
6. Treatment with any non-marketed investigational drug within 30 days prior to administration of [18F]-ML-10
7. Patient who received Whole Brain Radiation Therapy (WBRT) within 6 months prior screening and/or planned to receive WBRT 8 weeks post SRS
8. Patient receiving concurrent treatment with temozolamide or planned to receive temozolamide within 8 weeks post SRS
9. Woman of child-bearing potential who is not using an adequate and medically acceptable contraceptive method. Men who do not agree to use effective contraception during the study and for a period of 60 days following the last administration of [18F]-ML-10.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Assessment of the change in the uptake of [18F]-ML-10 by the target lesion(s) in response to SRS, as observed by comparing the PET/CT scans before and after SRS. Target lesion is defined as having a minimal diameter of 1.5 cm | 3 months

SECONDARY OUTCOMES:
Assessment of the relationship between the change in uptake of [18F]-ML-10 by the metastatic target lesions as observed in the PET/CT scans obtained before and after irradiation, and shrinkage of the metastatic target lesion, as assessed by MRI. | 3 months
Evaluation of the safety of [18F]-ML-10 when administered for 3 consecutive PET/CT scans to patients with brain metastases undergoing SRS. | one month

CONTACTS AND LOCATIONS:
Overall Officials: Yael Cohen, Study Director — Aposense Ltd.